CLINICAL TRIAL: NCT00006315
Title: Dose/Response of Exercise on Long Term Weight Loss
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 923; R01HL064991 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To examine the dose-response of exercise on long-term weight loss in overweight adult women.

DETAILED DESCRIPTION:
BACKGROUND:

Exercise is a key component of behavioral weight loss programs because of its effect on weight loss, body composition, cardiovascular disease risk factors, and other obesity related diseases such as type 2 diabetes mellitus. Despite these benefits, it is unclear whether there is an optimal exercise duration and/or intensity that will enhance long-term weight loss. The current public health recommendation for physical activity is for individuals to participate in at least 30 minutes of moderate intensity physical activity on most days of the week (approximately 150 minutes per week total). However, it is unclear whether this amount of exercise is adequate for long-term weight loss. Moreover, cross-sectional studies have shown that individuals that have been successful at long-term weight loss participate in levels of physical activity that are greater than the current public health recommendations.

DESIGN NARRATIVE:

The researchers hypothesized that adopting higher levels of exercise duration and/or intensity, coupled with a strong behavioral intervention would enhance long-term weight loss. To test this hypothesis, they recruited 200 overweight women and randomly assigned them to one of four treatment groups: (1) moderate intensity, moderate 1000cal/wk duration exercise, (2) vigorous intensity moderate duration exercise, (3) moderate 2000cal/wk intensity, high duration exercise, and (4) vigorous intensity, high duration exercise. All subjects participated in a 24-month behavioral weight loss program, with subjects attending group meetings and receiving periodic telephone contacts from the weight loss program, with subjects attending group meetings and receiving periodic telephone contacts from the interventionists. In addition, to facilitate the adoption of the exercise protocols, all subjects were provided with a home treadmill. Assessment of body weight occured at 0, 6, 12, and 24 months and exercise participation was measured throughout the program. In addition, body composition, cardiorespiratory fitness, cardiovascular disease risk factors, and mediators of behavior change were measured at 0, 6, 12, and 24 months.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Jakicic — University of Pittsburgh

REFERENCES:
- [Background] Jakicic JM, Wing RR, Winters-Hart C. Relationship of physical activity to eating behaviors and weight loss in women. Med Sci Sports Exerc. 2002 Oct;34(10):1653-9. doi: 10.1097/00005768-200210000-00018. PMID 12370568
- [Background] Jakicic JM, Gallagher KI. Exercise considerations for the sedentary, overweight adult. Exerc Sport Sci Rev. 2003 Apr;31(2):91-5. doi: 10.1097/00003677-200304000-00007. PMID 12715973
- [Background] Jakicic JM. The role of physical activity in prevention and treatment of body weight gain in adults. J Nutr. 2002 Dec;132(12):3826S-3829S. doi: 10.1093/jn/132.12.3826S. PMID 12468633
- [Background] Gallagher KI, Jakicic JM, Kiel DP, Page ML, Ferguson ES, Marcus BH. Impact of weight-cycling history on bone density in obese women. Obes Res. 2002 Sep;10(9):896-902. doi: 10.1038/oby.2002.123. PMID 12226138
- [Background] Jakicic JM, Marcus BH, Gallagher KI, Napolitano M, Lang W. Effect of exercise duration and intensity on weight loss in overweight, sedentary women: a randomized trial. JAMA. 2003 Sep 10;290(10):1323-30. doi: 10.1001/jama.290.10.1323. PMID 12966123
- [Derived] Jakicic JM, Marcus BH, Lang W, Janney C. Effect of exercise on 24-month weight loss maintenance in overweight women. Arch Intern Med. 2008 Jul 28;168(14):1550-9; discussion 1559-60. doi: 10.1001/archinte.168.14.1550. PMID 18663167